CLINICAL TRIAL: NCT03097562
Title: Wound Architecture and Functional Outcome After Cataract Surgery With Manual vs. Femtosecond Laser Assisted Procedures
Brief Title: Wound Architecture and Functional Outcome After Cataract Surgery With Manual vs.Femtosecond Laser Assisted Procedures
Acronym: CATALYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr. Paul Harasymowycz, Chief of Glaucoma Service University of Montreal, Maisonneuve-Rosemont Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: F11a-CEMTL-3355
Record Dates: First submitted 2016-06-10; First posted 2017-03-31 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Cataract
Keywords: Cataract; Femtosecond laser; Cornea; Anatomy; FSL; surgery
MeSH Terms: conditions — Cataract; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Post market study (Phase IV)
Masking Description: Consecutive patients who underwent cataract surgery using one of the following three types of surgical wound will be compared:
  1. Catalys - Initial wound parameters
  2. Catalys - Revised wound parameters
  3. Standard manual technique (MT control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT1 (Experimental): FLACS- Initial Wound parameters (CT1)
  Sample size calculation based on woundleak incidence estimated from preliminary results:
  * For CT1 vs MT, we will only need 10 per group to have 80% power assuming a 1:1 ratio of CT to MT and 5% type 1 error.
  * For CT1 vs CT2, we will need 22 per group to have 80% power (assuming 60% wound leakage in CT1 and 20% wound leakage in CT2, a 1:1 ratio, and a 5% type 1 error rate)
  * A total of 253 patients are eligible for this study, 101 with FLACS and 152 with Manual Cataract Surgery. We thus expect that our study population will allow adequate analysis of the main outcome parameters proposed herein.
  Interventions: Procedure: Femtosecond cataract surgery
- CT2 (Experimental): The revised profile CT2, consists of a wider anterior side cut angle (beveled corneal undercut) and a narrower posterior side cut angle compared to the initial CT1 profile. This new corneal incision profile is constructed to ensure a tigher wound closure and a better corneal wound reapposition.
  The traditional manual wound performed with a standard keratome wil be used as a reference.
  Interventions: Procedure: Femtosecond cataract surgery
- MT control group (Active Comparator): Standard manual technique (MT)
  Interventions: Procedure: Femtosecond cataract surgery

INTERVENTIONS:
Procedure: Femtosecond cataract surgery — Catalys create a circular opening for accessing and removing the cataract.
  Other Names: ReLACS

SUMMARY:
This study is the long term analysis of two types of FSL 3-plane corneal wound profiles, namely CT1 and CT2 obtained after a FSL cataract surgery.

DETAILED DESCRIPTION:
Femtosecond laser cataract surgery offers several major advantages for wound construction, including high precision, repeatability and a large variety of corneal wound profiles. The aim of this study is the long term analysis of two types of FSL 3-plane corneal wound profiles, namely CT1 and CT2, CT2 being constructed with a reversed front corneal incision segment to ensure tigher wound closure and better corneal wound reapposition. The traditional manual wound performed with a standard keratome will be used as a reference. As FSL cataract surgery may be associated with a greater incidence of wound leaks at the end of surgery as compared to manual wound construction with keratomes, this study will also aim at determining wich clinical and OCT wound parameters are associated with a higher likelihood of wound leaks.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive cases of cataract surgery performed between January 2015 and june 2015 by a single surgeon (PH) at the clinique d'ophtalmologie Bellevue, using either the Catalys or a manual technique.
* One eye per patient, the first eye
* Uneventful cataract only

Exclusion Criteria:

* Combined glaucoma filtering surgery
* Any previous corneal surgery in this eye
* Any pathology of the interior segment
* Inflammatory eye disease of the interior segment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1123 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Preservation of a physiological postoperative anatomy will be considered as a criterion of success | 2 Months
  Change in corneal anatomy as measured by the difference between pre-and postoperative corneal profile on OCT images

SECONDARY OUTCOMES:
The absence or a lower incidence of wound leak will also be considered as a criterion of success | 2 Months
  Presence or not of a wound leak necessitating a 10.0 Nylon to stop the leak

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harasymowycz, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Montreal Glaucoma Institut, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication of data and results in an Ophtalmology journal, conferences